CLINICAL TRIAL: NCT06381518
Title: Switching From Intravenous to Subcutaneous Infliximab in Adult Patients With Inflammatory Bowel Disease: Evaluation of Exposure Parameters
Brief Title: Switching From Intravenous to Subcutaneous Infliximab in Adult Patients With Inflammatory Bowel Disease
Acronym: SHUFFLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z2023165
Record Dates: First submitted 2024-03-12; First posted 2024-04-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: IBD; Infliximab; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is a prospective, single centre, open-label cohort study, conducted in Zuyderland Medical Centre in which adult IBD patients in remission on stable IV IFX therapy are switched to SC CT-P13 and is designed to compare the pharmacokinetics of SC CT-P13 to IV IFX and relate this to the pharmacodynamics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Infliximab monotherapy (Other): Adult patients (18-75 years old) on maintenance monotherapy of IV IFX.
  Interventions: Other: Switch to SC CT-P13.
- Cohort 2: infliximab combination therapy (Other): Adult patients on maintenance combination therapy of IV IFX with a thiopurine derivate or methotrexate.
  Interventions: Other: Switch to SC CT-P13.

INTERVENTIONS:
Other: Switch to SC CT-P13. — all patients in the study will switch from IFX to SC CT-P13

SUMMARY:
The aim of this study is to evaluate the IFX exposure (AUC), effectiveness, presence of ADAbs and treatment burden before and after switching from IV to SC IFX maintenance treatment in a real-world cohort of IBD patients with quiescent disease on IFX monotherapy and combination therapy of IFX and an immunomodulator.

Methods: this is a prospective, single centre, open-label cohort study, conducted in Zuyderland Medical Centre in which 36 adult IBD patients in remission on stable IV IFX therapy are switched to SC CT-P13 of which 18 patients use an immunomodulator in addition to IFX (cohort 2). After the switch to SC CT-P13, patients are followed for 24 weeks.

The study is subdivided into two phases: the IV IFX treatment phase before switching and the SC CT-P13 treatment phase after the switch. After enrolment, the subject receives a final dose of IV IFX according to their own maintenance schedule. Primary endpoints are the Area under the concentration-time curve (AUC) at steady state (1) before and after the switch to SC CT-P13 and (2) with or without concomitant immunomodulator during SC therapy. AUCs will be estimated using pharmacokinetic modelling in MwPharm. Besides IFX trough level, treatment related time expenditure, quality-of-life and patient satisfaction will be assessed before and after the switch.

DETAILED DESCRIPTION:
On demand.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years) with an confirmed diagnosis of IBD according to usual criteria, including previous endoscopic examination.
* Patients on IV IFX maintenance therapy at a stable dose and dosing interval for at least 16 weeks of 5-10 mg/kg every 6-8 weeks without side effects of IFX.
* IBD in clinical remission for at least 16 weeks without treatment with systemic corticosteroids in the previous 16 weeks. Clinical remission in adult patients is defined as a Harvey-Bradshaw index (HBI) < 4 for CD [18] or a partial Mayo Index (PMI) <2 for UC [19], with faecal calprotectin levels <250 μg/g faeces and CRP <10 mg/L.
* Concomitant immunomodulators are allowed, i.e. in stable doses were received for at least 12 weeks prior to study enrolment. These doses will be continued throughout the study, including azathioprine (AZA), 6-mercaptopurine (6-MP), tioguanine (TG) and MTX.
* Written informed consent

Exclusion Criteria:

* Patient <18 years of age.
* Allergy or hypersensitivity to any of the excipients of SC CT-P13.
* Patient with active perianal fistula.
* Patient with another autoimmune disease in addition to IBD.
* Patient treated concomitantly with another Mab in addition to IFX.
* Patients who, after starting IV IFX, have developed new contraindications to IFX according to European Public Assessment Report (EPAR).[3]
* Female patient who is currently pregnant or breastfeeding, or is planning to become pregnant or breastfeed within 6 months of the last dose of IFX.
* Patient has a serious acute or chronic medical or psychiatric condition that might increase the risk associated with study participation or investigational product administration or that might interfere with the interpretation of study results.
* Patients who, in the opinion of their general practitioner or investigator, should not participate in the study (e.g. non-adherence, mental health problems, illiteracy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) at steady state | 30-32 weeks
  AUC is estimated by pharmacokinetic modelling (MW Pharm)

SECONDARY OUTCOMES:
Quality of life score | 30-32 weeks
  Quality of life questionnaire (IBDQ-NL)
Patient satisfaction | 30-32 weeks
  5-points scale
Time expenditure | 30-32 weeks
  quationnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Sittard, Netherlands

IPD SHARING:
Plan to Share IPD: No